CLINICAL TRIAL: NCT06193577
Title: Single-centre, Prospective, Randomized, Placebo-controlled, Single-blind Clinical Trial to Evaluate the Efficacy of a Food Supplement Based on Phaseolus Vulgaris L. Dry Extract on the Modulation of Weight and Metabolic Parameters
Brief Title: Effect of Phaseolus Vulgaris L. Dry Extract on the Modulation of Weight and Metabolic Parameters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IBSA Farmaceutici Italia Srl (Industry)
Collaborators: Informapro Srl (Other); Universita degli Studi di Catania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IBSA-PHAS-0122
Record Dates: First submitted 2023-12-06; First posted 2024-01-05 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: Single-centre, prospective, randomized, placebo-controlled, single-blind clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phaseolus Vulgaris L. Dry Extract (Experimental): Test
  Interventions: Dietary Supplement: Phaseolus Vulgaris L. Dry Extract
- Placebo (Placebo Comparator): Control
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Phaseolus Vulgaris L. Dry Extract — Extracts of Phaseolus vulgaris (beans) in association with a balanced diet are known to reduce glycaemia and food intake in rodents and humans thus promoting weight loss.
  Arms: Phaseolus Vulgaris L. Dry Extract
Dietary Supplement: Placebo — The placebo control does not contain active ingredients.
  Arms: Placebo

SUMMARY:
Evaluation of the efficacy of Phaseolus vulgaris L. dry extract on weight modulation.

DETAILED DESCRIPTION:
Monocentric, prospective, randomized, single-blind clinical trial to evaluate the effects of Phaseolus vulgaris L. dry extract (test) on weight reduction and on metabolic parameters after 12 weeks of supplementation. The efficacy on weight reduction will be evaluated in comparison with the placebo group (control).

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged between 18 and 60 years
* BMI between 25 and 35 kg/m2
* Habitual consumption of three main meals a day
* Stable body weight during the 3 months prior to enrollment
* Commitment to adhere to the diet and avoid the use of other weight loss products during the study
* Commitment not to change lifestyle significantly for the entire duration of the study.
* Signing of informed consent

Exclusion Criteria:

* Hypergonadotropic hypogonadism and hypogonadotropic hypogonadism
* Diabetes mellitus
* Smoking > 10 cigarettes/day
* Alcohol > 2 alcohol units/day (equal to 24 g of ethanol)
* History of eating disorders during the 12 months prior to enrollment
* Use of any drug or product to treat obesity (e.g. meal replacements)
* Presence of acute or chronic gastrointestinal diseases
* Active use of drugs that could influence the functions: gastrointestinal (e.g. laxatives, etc.), insulin (insulin sensitizers, etc.) and/or testicular (hormones, substances that influece testosterone production
* Known sensitivity to the ingredients of the preparation
* Any other clinical condition judged by the investigator to be incompatible with participation in the trial

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in weight | 0, 12 weeks
  Weight evaluation before and after treatment

SECONDARY OUTCOMES:
Change in weight | 0, 4, 8, 18 weeks
  Weight evaluation before and after treatment
Change in Body Mass Index | 0, 4, 8, 12, 18 weeks
  BMI evaluation before and after treatment
Change in glycemia | 0, 4, 8, 12, 18 weeks
  Glycemia evaluation before and after treatment
Change in total testosterone levels | 0, 4, 8, 12, 18 weeks
  Total testosterone levels evaluation before and after treatment
Change in LH levels | 0, 4, 8, 12, 18 weeks
  Luteinizing hormone (LH) levels evaluation before and after treatment
Change in FSH levels | 0, 4, 8, 12, 18 weeks
  Follicle-stimulating hormone (FSH) levels evaluation before and after treatment
Change in SHBG levels | 0, 4, 8, 12, 18 weeks
  Sex Hormone Binding Globulin (SHBG) levels evaluation before and after treatment
Change in 17-beta-estradiol levels | 0, 4, 8, 12, 18 weeks
  17-beta-estradiol levels evaluation before and after treatment
Change in insulin levels | 0, 4, 8, 12, 18 weeks
  Insulin levels evaluation before and after treatment
Change in albumin levels | 0, 4, 8, 12, 18 weeks
  Albumin levels evaluation before and after treatment
Change in carboxylated osteocalcin (cxOCN) levels | 0, 4, 8, 12, 18 weeks
  Carboxylated osteocalcin levels evaluation before and after treatment
Change in uncarboxylated osteocalcin (ucOCN) levels | 0, 4, 8, 12, 18 weeks
  Uncarboxylated osteocalcin levels evaluation before and after treatment
Change in calculated free testosterone (CFT) concentrations | 0, 4, 8, 12, 18 weeks
  Calculated free testosterone (CFT) concentrations evaluation before and after treatment
Sperm count | 0, 12, 18 weeks
  Sperm count before and after treatment
Sperm motility | 0, 12, 18 weeks
  Sperm motility before and after treatment
Sperm morphology evaluation | 0, 12, 18 weeks
  Sperm morphology evaluation before and after treatment
Sperm vitality | 0, 12, 18 weeks
  Sperm vitality evaluation before and after treatment
Tunel test | 0, 12, 18 weeks
  Sperm DNA fragmentation evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Calogero, Prof., Principal Investigator — Università di Catania
Locations (1):
- A.O.U. Policlinico "G. Rodolico - San Marco", Catania, Catania, Italy